CLINICAL TRIAL: NCT00511472
Title: A Multicenter, 2-Part, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-0941 on Postprandial Plasma Glucose Concentrations After Daily Administration MK-0941 Before Each Meal (q.a.c) in Subjects With Type 2 Diabetes Being Treated With Basal Insulin
Brief Title: An Investigational Drug Study in Adults With Type 2 Diabetes on Basal Insulin (MK-0941-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-006; 2007_596; MK-0941-006
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Results first posted 2012-07-11 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MK-0941 (Experimental)
  Interventions: Drug: MK-0941; Drug: LANTUS insulin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: LANTUS insulin

INTERVENTIONS:
Drug: MK-0941 — In Titration Scheme #1, MK-0941/matching placebo was initiated at 10-mg q.a.c. dose and increased on a daily basis (Titration Dose [TD] Days 1 to 4 of the Titration Phase 1) in 10-mg q.a.c. increments.
  Titration Scheme #2 was a flexible-dose titration scheme in which MK-0941/matching placebo was given at a dose determined by a pre-prandial plasma glucose concentration for the subsequent meal on the previous day of administration on Days 1 to 4 of the Titration Phase 2.
  Arms: MK-0941
Drug: Placebo — 10 mg Placebo (Pbo), 20 mg Pbo, 30 mg Pbo or 40 mg Pbo q.a.c.
  Arms: Placebo
Drug: LANTUS insulin — LANTUS insulin dose will be similar to participant's previous dose of immediate or long-acting insulin
  Other Names: LANTUS

SUMMARY:
A study to assess safety, pharmacokinetics (PK), and pharmacodynamics (PD) of MK-0941 in Type 2 diabetics being treated with basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-childbearing potential) between 18 to 70 years of age
* Diagnosed with Type 2 Diabetes and currently being treated with basal insulin
* Smokers may participate, but they are limited to 10 cigarettes per day while at the clinic and must follow clinic smoking rules

Exclusion Criteria:

* History of Type 1 diabetes
* Treated with peroxisome proliferator-activated receptor (PPAR) agonists within 12 weeks prior to study start
* History of severe hypoglycemia
* Allergic to insulin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941: Participants receiving multiple daily before each meal (q.a.c.) administrations of MK-0941 while on basal insulin.
- Placebo: Participants receiving placebo while on basal insulin.
Period: Overall Study
Arm/Group | MK-0941 | Placebo
Started | 47 | 23
Completed | 44 | 17
Not Completed | 3 | 6
Not completed — Clinical Adverse Event | 1 | 2
Not completed — Laboratory Adverse Event | 0 | 2
Not completed — Not reported | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0941 | Placebo | Total
Number analyzed (Participants) | 47 | 23 | 70
Age, Customized [Number; unit: participants]
  <22 years | 0 | 0 | 0
  22 to 69 years | 47 | 23 | 70
  >69 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 28 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event During the Study
Time Frame: 39 days
Population: All participants who experienced one or more adverse events during the study
Measure: Number; unit: participants
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 47 | 23
participants | 46 | 21

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event - Titration Scheme 1
Description: In Titration Scheme #1, MK-0941/matching placebo was initiated at 10-mg q.a.c. dose and increased on a daily basis in 10-mg q.a.c. increments on Titration Dose [TD] Days 1 to 4 of the Titration Phase 1 of the study.
Time Frame: 25 days
Population: All participants who experienced one or more adverse events within 25 days of Titration Scheme 1
Measure: Number; unit: participants
Groups:
- MK-0941: Participants receiving multiple daily before each meal (q.a.c.) administrations of MK-0941 according to Titration Scheme #1 while on basal insulin.
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 23 | 12
participants | 20 | 11

3. Secondary Outcome: Number of Participants Who Experienced an Adverse Event - Titration Scheme 2
Description: Titration Scheme #2 (Titration Phase, Days 1 to 4) was a flexible-dose titration scheme in which MK-0941/matching placebo was given at a dose determined by a pre-prandial plasma glucose concentration for the subsequent meal on the previous day of administration.
Time Frame: 25 days
Population: All participants who experienced one or more adverse events within 25 days of Titration Scheme 2
Measure: Number; unit: participants
Groups:
- MK-0941: Participants receiving multiple daily before each meal (q.a.c.) administrations of MK-0941 according to Titration Scheme #2 while on basal insulin.
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 24 | 11
participants | 22 | 10

4. Secondary Outcome: 24-Hour Weighted Mean Blood Glucose Levels (mg/dL) by Treatment Group on Day 7
Description: Measurement of the 24-hour weighted mean blood glucose levels of participants receiving MK-0941 or placebo while on basal insulin on Day 7.
Time Frame: 24 hours
Population: All participants who had 24-hour weighted mean blood glucose levels evaluated on Day 7
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Groups:
- MK-0941 (Titration Group 1): Participants receiving multiple daily before each meal (q.a.c.) administrations of MK-0941 according to Titration Scheme #1 while on basal insulin.
- MK-0941 (Titration Group 2): Participants receiving multiple daily before each meal (q.a.c.) administrations of MK-0941 according to Titration Scheme #2 while on basal insulin.
Arm/Group | MK-0941 (Titration Group 1) | MK-0941 (Titration Group 2) | Placebo
Number analyzed (Participants) | 22 | 24 | 20
mg/dL | 155.5 (62.9) | 151.3 (47.4) | 201.6 (54.9)
Statistical Analysis 1: Comparison: MK-0941 (Titration Group 1) vs Placebo; For the least square mean difference - baseline in the ANOVA model = glucose value at Titration Day 1 pre-Breakfast for Titration Group 1; Test type: Superiority or Other; p = 0.001, ANOVA; Mean Difference (Final Values) = 46.10, 90% CI 2-sided [22.71 to 69.50], Standard Error of Mean 14.15
Statistical Analysis 2: Comparison: MK-0941 (Titration Group 2) vs Placebo; For the least square mean difference - baseline in the ANOVA model = glucose value at Titration Day 1 pre-breakfast for Titration Group 2; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 50.28, 90% CI 2-sided [27.68 to 72.88], Standard Error of Mean 13.67

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event During the Outpatient Treatment Period
Description: During the Outpatient Treatment Period, participants were followed for an additional 2 weeks while at home.
Time Frame: Outpatient Days 1 to 14
Population: All participants who experienced one or more adverse events during the Outpatient Treatment Period.
Measure: Number; unit: participants
Groups:
- MK-0941: Participants receiving individualized doses of MK-0941 while on basal insulin
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 44 | 17
participants | 20 | 11

ADVERSE EVENTS:
Time Frame: 25 days
Description: All participants who received at least 1 dose of study drug
Groups:
- MK-0941 Titration 1: Participants receiving multiple daily q.a.c. administrations of MK-0941 according to Titration Scheme 1 while on basal insulin.
- MK-0941 Titration 2: Participants receiving multiple daily q.a.c. administrations of MK-0941 according to Titration Scheme 2 while on basal insulin.
- Placebo Titration 1; Placebo Titration 2: Participants receiving placebo while on basal insulin.
Arm/Group | MK-0941 Titration 1 | MK-0941 Titration 2 | Placebo Titration 1 | Placebo Titration 2
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/24 | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 20/23 | 21/24 | 11/12 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0941 Titration 1 (N=23) | MK-0941 Titration 2 (N=24) | Placebo Titration 1 (N=12) | Placebo Titration 2 (N=11)
Multiple Injuries (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0941 Titration 1 (N=23) | MK-0941 Titration 2 (N=24) | Placebo Titration 1 (N=12) | Placebo Titration 2 (N=11)
Dry Eye (Eye disorders) | 1 | 2 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 5 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 7 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 2 | 0
Headache (Nervous system disorders) | 9 | 10 | 5 | 6
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 2
Tremor (Nervous system disorders) | 4 | 2 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 1 | 1 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Vessel Puncture Site Pain (General disorders) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Peripheral Coldness (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.